CLINICAL TRIAL: NCT05464563
Title: Study by Electroencephalography of the Link Between the Lack of Self-compassion and the Disorder of Empathy in Schizophrenia
Acronym: SCE-SCHIZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A01913-38
Record Dates: First submitted 2022-04-21; First posted 2022-07-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Patients have electroencephalogram records during :
  * a phase of rest;
  * a task of self-compassion
  * a task of empathy.
  Interventions: Device: Electroencephalogram
- Control group (Experimental): Healthy volunteers have electroencephalogram records during :
  * a phase of rest;
  * a task of self-compassion
  * a task of empathy.
  Interventions: Device: Electroencephalogram

INTERVENTIONS:
Device: Electroencephalogram — An electroencephalogram is recorded during a task of rest then self-compassion and then empathy.

SUMMARY:
This research project focuses on a fundamental element of the psychopathology of schizophrenia, that is to say, the disorders of self-awareness and on the functional alterations associated with it, that is to say, self-compassion deficit and empathy disorder.

It will be a question of better understanding the neuro-functional mechanisms which underlie the lack of self-compassion and the disorder of empathy in schizophrenia, the relationship that these disorders maintain between them but also the relationship that they maintain with the general psychopathology of schizophrenia and, in particular, with the abnormalities of the self. In other words, the overall framework of this project is that of the link between the psychopathology of schizophrenia and the functional impairment associated with it. Its specific field of application is that of the link between self-awareness disorders, self-compassion deficit and empathy disorder. For this, this project proposes a methodological approach combining the recording of intrinsic and extrinsic brain activity using high-density electroencephalography (EEG).

DETAILED DESCRIPTION:
This study includes patients (n=30) and healthy volunteers (n=30).

At inclusion visit, participants have:

* a psychiatric evaluation;
* self evaluation of: empathy, self-compassion, émotionnel processing, anxiety, insight, perceptual aberration and quality of life;
* training to practise of self-compassion and empathy (for patients only).

During the phase of experimentation, the participants have electroencephalogram exams during a rest phase, a self-compasion task and an empathy task.

ELIGIBILITY:
Inclusion Criteria for the patient group :

* patients with a schizophrenic or schizoaffective disorder according to the DSM-5 criteria (axis 1), with no other pathology of axis 1, except addiction to tobacco
* patients stabilized for at least 3 months for their psychotic disorders
* patients with disease duration > 2 years but < 20 years
* patients whose treatment has not been changed or modified in the previous month
* patients on stable treatments who should not change treatment during the study (good compliance, good tolerance)
* patients who do not benefit from a neuromodulation protocol for their symptoms (rTMS, TDCS)
* patients who do not benefit from a cognitive remediation program
* patients between the ages of 18 and 60
* men and women
* patients with normal or corrected vision
* patients without mental impairment
* patients without neurological impairment (epilepsy, encephalopathy, head trauma)
* patients with a sufficient command of French
* patients free or under protective measures
* patients benefiting from coverage by a social security scheme or benefiting from it through a third party
* Having given their consent to participate in the study after having received written, clear and fair information (and after obtaining the consent of the tutor/curator if applicable)

Exclusion Criteria for the patient group :

* patients with an axis 1 pathology other than a schizophrenic or schizoaffective disorder (in particular, psychic trauma revealed by MINI and symptoms of PTSD (current as lifetime))
* patients with an addiction to alcohol or other toxic substances, except tobacco
* patients with suicidal intentionality
* patients not stabilized for their psychotic disorders and with regard to their antipsychotic treatments
* patients receiving antiepileptic treatment with mood-regulating, antidepressant and anxiolytic properties
* patients receiving benzodiazepine treatment that they could not stop 72 hours before the EEG
* patients with disease duration < 2 years or > 20 years
* patients with an IQ < 70
* patients benefiting from a neuromodulation protocol (rTMS, TDCS)
* patients benefiting from a cognitive remediation program
* patients with a PANSS > or = 5 for items G8 (hostility) and P7 (non-cooperation)
* patients aged < 18 years or > 60 years
* patients with mental impairment
* patients with neurological impairment (epilepsy, encephalopathy, head trauma)
* patients with documented neurological pathology or medical condition that may explain the psychotic manifestations
* patients who do not speak French well enough
* subjects residing within a radius greater than 50 km from the hospital
* patients hospitalized under duress
* patients without social security

Inclusion Criteria for the control group:

* healthy volunteers without schizophrenic or schizoaffective disorder and without other psychiatric pathologies as defined by the DSM 5 (axis 1) (in particular, absence of psychic trauma revealed by the MINI and of PTSD (current as whole life))
* subjects aged 18 to 60
* men and women
* subjects with normal or corrected vision
* subjects without mental impairment
* subjects without neurological impairment (epilepsy, encephalopathy, head trauma)
* free subjects, without guardianship or curatorship or subordination
* subjects benefiting from coverage by a social security scheme or benefiting from it through a third party
* Having given their consent to participate in the study after having received written, clear and honest information.

Exclusion Criteria for the control group:

* subjects with a psychiatric pathology as defined in the DSM-5 (axis 1) (in particular, psychic trauma revealed by the MINI and symptoms of PTSD (current as lifetime))
* subjects aged < 18 years or > 60 years
* subjects with a mental deficiency
* subjects with neurological pathology
* subjects with a medical condition preventing them from participating in the study
* subjects residing within a radius greater than 50 km from the hospital
* subjects under guardianship or curatorship
* subjects not benefiting from a Social Security scheme or not benefiting from it through a third party

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the temporal parameters of the EEG microstates C, D, E and F (duration, contribution, occurrence) and the inter-subject correlation index during the practice of self-compassion and the practice of empathy. | through study completion, an average of 36 months.
  Correlation between the temporal parameters of the EEG microstates C, D, E and F (duration, contribution, occurrence) and the inter-subject correlation index during the practice of self-compassion and the practice of empathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No